CLINICAL TRIAL: NCT05353452
Title: Collaborative Care for Anxiety and Depression in Posttraumatic Epilepsy
Brief Title: Collaborative Care in Posttraumatic Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00084191; 40010222 (Other: Department of Defense); CDMRP-EP210036 (Other: CDMRP)
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Epilepsy, Post-Traumatic
Keywords: epilepsy; neurological care; collaborative care; anxiety; depression
MeSH Terms: conditions — Epilepsy, Post-Traumatic; Epilepsy; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Care (Experimental): Participants in this arm will receive 24 weeks of neurology based collaborative care.
  Interventions: Behavioral: Neurology Based Collaborative Care
- Standard of Care (SOC) (Active Comparator): Participants in this arm will receive provider-recommended clinic visits, prescriptions, testing, and referrals.
  Interventions: Behavioral: SOC Neurological care

INTERVENTIONS:
Behavioral: Neurology Based Collaborative Care — Twenty-four week, evidence-based remote collaborative care model initiated around the time of a neurology visit. The collaborative care team roles include the care manager, psychiatrist, and psychologist/social worker who interact with the patient participant and the patient's neurologist.
  Arms: Collaborative Care
Behavioral: SOC Neurological care — Usual neurology care means ongoing, epilepsy provider-recommended clinic visits, prescriptions, testing and referrals from their epilepsy provider. Mental health referrals or prescribing of antidepressants may potentially occur in this group; these types of interventions will be tracked at outcome assessments.
  Arms: Standard of Care (SOC)

SUMMARY:
The purpose of this research is to evaluate a 6 month change in quality of life in subjects who receive collaborative care calls compared to those subjects who receive usual neurology care. This is a 2-site trial comparing a 24 week neurology-based collaborative care program to usual neurology care among a total of 60 adults with post-traumatic epilepsy.

DETAILED DESCRIPTION:
The study will compare collaborative care versus usual care among N=60 adults with post-traumatic epilepsy and anxiety and/or depression symptoms in Veterans Administration (N=20) and civilian university (N=40) settings at the Salisbury VA and Atrium Health Neurology. This single-blind study will evaluate effectiveness and implementation of a remotely-delivered, 24-week team-delivered collaborative care intervention, with features adapted from VA Primary Care Mental Health Integration and Whole Health, as well as an existing Family Medicine Collaborative Care Program at AHWFB.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures
* Diagnosis of post-traumatic epilepsy, defined by the following:

  1. Epilepsy diagnosis based on neurology clinician impression of diagnosis or electroencephalogram (EEG) findings (EEG findings: presence of interictal epileptiform discharges on EEG or ictal EEG recording of seizure definitively documenting epilepsy diagnosis)
  2. History of at least mild traumatic brain injury based on the MIRECC (Mental Illness Research, Education, and Clinical Center) TBI (Traumatic Brain Injury) screening instrument or verified TBI history based on MIRECC research database
  3. TBI pre-dated onset of epilepsy (NINDS post-traumatic epilepsy screening form)
* Anxiety or depression symptoms--Generalized Anxiety Disorder scale (GAD-7) ≥8 or Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) >13
* Receiving clinical neurological care at one of the study sites

Exclusion Criteria:

* Active ongoing treatment by a psychiatrist without the potential to benefit from additional collaborative care for anxiety or depression in the judgement of the investigators
* Active suicidal ideation
* History of past suicide attempt
* Unstable drug or alcohol abuse
* Unstable or progressive comorbid medical condition
* Current participation in another treatment or intervention study
* Cognitive limitations precluding completion of anxiety and depression self-report instruments on paper, electronically, or by interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Emotional Subscale-Change in Quality of Life in Epilepsy-31(QOLIE-31) | Baseline through Month 6
  This is a clinically meaningful patient reported outcome measure that was demonstrated to improve in collaborative care efficacy trials in distinct patient groups (including with various different types of medical illness) Score ranges from 0-100 with higher score indicating better quality of life

SECONDARY OUTCOMES:
Subject Adherence to Intervention | Week 12
  Proportion of intervention arm participants who attend 50% or more of the care management calls in the first 12 weeks of the intervention.
Change in Epilepsy specific QOLIE-31 score | Baseline through Month 6
  Score ranges from 0-100 with higher score indicating better epilepsy-specific quality of life.
Change in Beck Depression Inventory-II (BDI-II) score | From baseline through Month 6
  Depression symptom questionnaire-score ranges from 0-61, with higher score indicating more severe depression symptoms.
Change in Beck Anxiety Index (BAI) score | From baseline through Month 6
  Anxiety symptom questionnaire-score ranges from 0-61, with higher score indicating more severe anxiety symptoms.

OTHER OUTCOMES:
Feasibility of Intervention Measure (FIM)-Subject Perspective | Baseline and Month 3
  Questionnaire to help determine feasibility of collaborative care from participants' perspectives. Score ranges from 5 to 20, with higher score indicating greater feasibility.
FIM-Neurologist Perspective | Baseline and Month 3
  Questionnaire to help determine feasibility of collaborative care from neurologists' perspectives. Score ranges from 5 to 20, with higher score indicating greater feasibility.
Acceptability of Intervention Measure (AIM)-Subject Perspective | Baseline and Month 3
  Questionnaire to help determine acceptability of collaborative care from participants' perspectives. Score ranges from 5 to 20, with higher score indicating greater acceptability.
AIM-Neurologist Perspective | Baseline and Month 3
  Questionnaire to help determine acceptability of collaborative care from neurologists' perspectives. Score ranges from 5 to 20, with higher score indicating greater acceptability.
Intervention Appropriateness Measure (IAM)-Subject Perspective | Baseline and Month 3
  Questionnaire to help determine appropriateness of collaborative care from participants' perspectives. Score ranges from 5 to 20, with higher s indicating greater appropriateness.
IAM-Neurologist Perspective | Baseline and Month 3
  Questionnaire to help determine appropriateness of collaborative care from neurologists' perspectives. Score ranges from 5 to 20, with higher score indicating greater appropriateness.
Proportion of participants who attend at least 50% of Scheduled Calls | Week 12 and Week 24
  Pertains only to participants randomized to collaborative care intervention
Individual Participant Collaborative Care Call Attendance Percentage | Week 12 and Week 24
Seizure Frequency | Baseline, Month 3, and Month 6
  Number of seizures experienced by participants
Change in BDI-II Score | From Baseline through Month 3
  Depression symptom questionnaire-score ranges from 0-61, with higher score indicating more severe depression symptoms.
Change in BAI Score | From Baseline through Month 3
  Anxiety symptom questionnaire- score ranges from 0-61, with higher score indicating more severe anxiety symptoms.
Change in Epilepsy specific QOLIE-31 Score | From Baseline through Month 3
  Score ranges from 0-100 with higher scores indicating better epilepsy-specific quality of life.
Emotional Subscale-Change in QOLIE-31 Score | Baseline through Month 3
  This is a clinically meaningful patient reported outcome measure that was demonstrated to improve in collaborative care efficacy trials in distinct patient groups (including with various different types of medical illness) Score ranges from 0-100 with higher score indicating better quality of life.
Change in Neurological Disorders Depression Inventory-Epilepsy (NDDI-E) | From Baseline through Month 6
  Depression symptom questionnaire specifically for those with epilepsy-score ranges from 6 to 24, with a score >15 indicating presence of a likely major depressive episode.
Change in Mini International Psychiatric Interview (MINI) | From Baseline through Month 6
  Validated diagnostic interview for Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-V) psychiatric diagnoses. The instrument indicates whether a current diagnosis of a DSM-V mood or anxiety disorder is present. This outcome will assess for change in presence of a current anxiety or depressive disorder at 6-months compared to baseline.
Change in Generic Quality of Life-SF-36 | From Baseline through Month 6
  This instrument is composed of 8 subscales, each calculated separately on a scale of 0-100, with higher score indicating better generic health-related quality of life for that subscale. This exploratory outcome pertains to the following subscales: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning.
Change in Liverpool Seizure Severity Scale (LSSS) | From Baseline through Month 6
  Seizure severity questionnaire- score ranges from 0 to 100, with higher score indicating increased seizure severity.
Prescription Adherence | Month 6
  Collected via review of pharmacy refills--number expected divided by number taken.
Change in Liverpool Adverse Effect Profile (LAEP) | From Baseline through Month 6
  Adverse effect questionnaire-score ranges from 19 to 76, with higher score indicating greater burden of adverse effects.
Change in Generalized Anxiety Disorders- 7(GAD-7) Score | From Baseline through month 3, From Baseline through month 6
  Questionnaire measuring anxiety symptoms-score ranges from 0 to 21, with higher score indicating increased anxiety symptoms.
Change in Patient Health Questionnaire-9 (PHQ-9) Score | From Baseline through month 3, From Baseline through month 6
  Score ranges from 0 to 27, with higher score indicating increased depression symptoms.
Emergency Department (ED)/Hospitalization Visits | From baseline through Month 6
  Number of hospitalizations or visits to ED.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi M. Munger Clary, MD, MPH, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munger Clary HM, Snively BM, Cagle C, Kennerly R, Kimball JN, Alexander HB, Brenes GA, Moore JB, Hurley RA. Collaborative Care to Improve Quality of Life for Anxiety and Depression in Posttraumatic Epilepsy (CoCarePTE): Protocol for a Randomized Hybrid Effectiveness-Implementation Trial. JMIR Res Protoc. 2024 Nov 13;13:e59329. doi: 10.2196/59329. PMID 39535875